CLINICAL TRIAL: NCT06395129
Title: Implementing a Low Dead-space Injecting Equipment Distribution Program for People Who Inject Drugs in Low- and Middle-income Countries: a Process and Outcome Evaluation
Brief Title: Low Dead-space Injecting Equipment Distribution Program for People Who Inject Drugs in Low- and Middle-income Countries
Status: Recruiting | Type: Observational
Sponsor: Médecins du Monde (Other)
Collaborators: UNITAID (Other); Burnet Institute (Other); International Network of People who Use Drugs (Unknown); University of Bristol (Other); Frontline AIDS (Other); Caritas (Unknown); Drug-free and preventitve healthcare organisation Nigeria (Unknown); National Viral Hepatitis and STI Control Program Nigeria (Unknown); PATH (Other); Population Services International (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: HepC LDSS
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Drug Use; Hepatitis; Hiv
Keywords: Low dead-space needles and syringes; Qualitative interviews; LDSS/N; High dead space needles/syringes (HDSS/N); Rapid diagnostic test (RDT); Feasibility; Acceptability; Cost effectiveness; Modelling; Focus group discussions; Harm Reduction; Values and preferences; Needle and syringe exchange program; Blood borne virus
MeSH Terms: conditions — Hepatitis; Acquired Immunodeficiency Syndrome; Harm Reduction | interventions — Needles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cohort study: All participants in the cohort study will undergo surveys, HIV, and HCV testing at four possible timepoints (baseline, 6-months, 12-months, and if time permits 18-months).
  They will also have access to the study sites usual services, and the introduced LDSS/N.
  Interventions: Device: Low dead-space syringes/needles; Device: Hepatitis C Antibody Rapid Diagnostic Test; Device: HIV rapid Diagnostic Test

INTERVENTIONS:
Device: Low dead-space syringes/needles — LDSS/N are a type of syringe/needle which retains less residual blood following an injecting event when compared to HDSS/N.
  Other Names: LDSS/N
Device: Hepatitis C Antibody Rapid Diagnostic Test — Administered up to 4 times, at baseline, 6-months, 12-months, and 18-months
  Other Names: HCV RDT
Device: HIV rapid Diagnostic Test — Administered up to 4 times, at baseline, 6-months, 12-months, and 18-months
  Other Names: HIV RDT

SUMMARY:
Implementation and evaluation of a distribution program for low dead-space syringes/needles (LDSS/N) in Armenia, Georgia, and Tanzania, Egypt, Nigeria, Vietnam, India, Ukraine, and South Africa. This study aims to generate evidence on best practice LDSS/N distribution programs which will enhance acceptability and sustain high levels of LDSS/N uptake.

People who inject drugs and access needle and syringe programs will be invited to attend up to three focus group discussion rounds (with 25 participants in each focus group round) to inform and provide feedback on a concurrent distribution program of LDSS/N.

Throughout distribution, a cohort study will be run alongside distribution with 240 participants enrolled per country (with the exception of Nigeria, where 480 participants will be recruited) who will undergo HIV and HCV testing and answer surveys on their sociodemographic and behavioral status. Key informant interviews will also be held with participating staff and stakeholders to evaluate the feasibility and acceptability of this program.

Primary outcomes assessed through this study include 1) community values and preferences for LDSS/N, 2) barriers and facilitators to accessing LDSS/N, 3) feasibility and effectiveness of the distribution program on increasing LDSS/N uptake, 4) model the potential public health impact and cost effectiveness of LDSS/N distribution in this setting.

DETAILED DESCRIPTION:
This study will recruit people who inject drugs to inform and evaluate the selection and distribution of low dead-space needles and syringes (LDSS/N) at their existing NSP services.

The interventions include: low- dead-space needles and syringes; and knowledge mobilisation through Focus Group Discussions (FGDs) and peer education.

Specifically, in Phase 1, people who inject drugs will be recruited at each study site to participate in FGDs, in which they will be presented with a selection of new LDSS/N products, provided information about their advantages regarding blood borne virus (BBV) transmission risk, and invited to discuss their values and preferences regarding needle- and syringe choice to inform the selection of LDSS/N to be piloted for scaled up distribution at their study sites.

Following the FGDs, during Phase 2 people who inject drugs who are registered clients at participating NSP services can enroll in a 6-week pilot period during which they will have access to a small selection of new LDSS/N products alongside the usual services they access at the study site or needle and syringe program (NSP). When the 6 week pilot phase concludes, participants will be invited to participate in a second round of FGDs, where they will be asked reflect on their experiences using the new LDSS/N products and share their opinions on which products to select for scaled up distribution to all clients accessing the study sites.

In Phase 3, a small selection LDSS/N (2-5) will be made available alongside the usual needles- and syringes and other existing harm reduction services at the study site/NSPs. During this period, two forms of data will be collected, 1) routine programmatic data, and 2) data from a concurrent cohort study.

The routine programmatic data collected will include information already routinely collected by the sites when individuals attend (site specific client ID, type and quantity of needles/syringes (N/S) collected) along with two additional questions 'Did you use a LDSS/N the last time you injected?" and "Thinking about the last week, for how many of your injections did you use a LDSS/N?'. No identifiable data will be recorded as part of routine programmatic data collection, therefore individuals included in this process are not considered 'participants' and will not undergo informed consent. This data will be used for the purposes of monitoring and evaluating LDSS/N uptake.

Alongside this distribution period, 240 people per country who inject drugs accessing participating study sites will be recruited into an observational cohort study. Participants will be asked to undergo HIV and HCV antibody testing and to answer surveys on demographic and behavioral activities at four timepoints (baseline, 6-months, 12-months, 18-months).

At the conclusion of the distribution period, a third round of FGDs will be run to assess the acceptability and impact of the LDSS/N distribution program. Key informant interviews with study staff and key stakeholders will also be completed to explore the feasibility and effectiveness of the LDSS/N program.

Following all data collection, mathematical modelling will estimate the impact and cost-effectiveness of scaling up LDSS/N for people who inject drugs at a country-level, including modelling the impact on BBV transmission.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years (note that country-specific protocols may include participants aged ≥16 where appropriate and relevant);
* Reporting a history of recent (past month) injection drug use;
* Accessing the NSP to receive injecting equipment at either a facility, mobile service or through outreach and have an accompanying assigned program unique ID;
* Able to understand and communicate in the local language(s);
* If self-reporting HCV/HIV negative status, interested in and agreeing to undergo HCV and HIV testing; and
* Willing and able to provide informed consent to take part in the study.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study sites will set a target for participation among women in line with the percentage of women accessing needle/syringe programmed locally. Where data is not currently available on gender, or if attendance is very low, the investigators will aim to recruit a minimum quota of 15% to ensure meaningful participation among women.
Study Population: People aged 18+ who report injecting drug use
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a community values and preferences informed LDSS/N distribution program on increasing LDSS uptake among people who inject drugs | 18 months
  Defined as reported exclusive use of LDSS/N vs not exclusive use of LDSS/N

SECONDARY OUTCOMES:
Understanding community values and preferences for LDSS/N in the context of other harm reduction supplies available to people who inject drugs | 18 months
  Identified through focus group discussions
Barriers and facilitators to access and uptake of LDSS/N among people who inject drugs | 18 months
  Assessed through surveys and focus group discussions
Differences in blood borne virus (HIV/HCV) incidence between those who exclusively use LDSS/N and those who do not | 18 months
Model the potential public health impact (HCV and HIV infections averted) and cost-effectiveness of LDSS/N distribution for people who inject drugs within harm reduction settings | 18 months
Identifying the enablers and challenges affecting the supply chain for LDSS/N | 18 months
Document the legal, social, and regularity enablers and challenges affecting the successful introduction and maintenance of LDSS/N distribution | 18 months
Evaluate LDSS/N demand creation approaches | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stoové, Principal Investigator — Burnet
Locations (9):
- Real World Real People, Yerevan, Armenia
- Georgia (3):
  - Step to Future, Gori
  - New Vector, Rustavi
  - Hepa+, Tbilisi
- Tanzania (5):
  - Mukikute, Dar es Salaam
  - Peer 2 Peer, Dar es Salaam
  - Yovaribe, Ilala
  - Mefada, Kinondoni
  - STEPS Tanzania, Ubungo

IPD SHARING:
Plan to Share IPD: Undecided